CLINICAL TRIAL: NCT02058511
Title: Intraoperative Use of Infrared Pupillometry During General Anesthesia to Predict Pain and Quality of Regional Anesthesia After Surgery
Brief Title: Infrared Pupillometry During General Anesthesia to Predict Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Preliminary results showed no ability to predict pain by measuring hippus with pupillometry
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Matthias Behrends, Associate Clinical Professor, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pupillometry and Analgesia
Record Dates: First submitted 2014-02-04; First posted 2014-02-10 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Postoperative Pain; Objective Assessment of Sedation
MeSH Terms: conditions — Pain, Postoperative | interventions — Neoadjuvant Therapy; Maintenance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention Group (Experimental): all enrolled patients undergo the same protocol/ treatment:
  Anesthesia Premedication, Induction and Maintenance Pupillometry after administration of anesthetic drugs
  Interventions: Drug: Anesthesia Premedication, Induction and Maintenance; Procedure: Pupillometry after administration of anesthetic drugs

INTERVENTIONS:
Drug: Anesthesia Premedication, Induction and Maintenance — The enrolled patients receive standard of care general anesthesia for knee arthroscopy. No additional pharmacological interventions are performed in study participants.
  The administered drugs, as outlined in the arms section, are midazolam, fentanyl, propofol, and sevoflurane. Study patients receive analgesic drugs as needed in the recovery room if they experience pain.
Procedure: Pupillometry after administration of anesthetic drugs — All study patients receive the standard of anesthetic care. Every time a anesthetic drug has been administered, changes in pupillary oscillations will be recorded.
  Assessment of pupil size and movements by shining infrared light into the eye and measuring the reflection over a 20 s period
  The administered drugs are:
  Midazolam 1-2 mg iv, Fentanyl 1mcg/kg body weight, Propofol for anesthesia induction 2-2.5 mg/kg body weight, Sevoflurane as needed for maintenance of general anesthesia.

SUMMARY:
The study comprises of a series of pupillary measurements using infrared pupillometry in patients undergoing arthroscopic knee surgery of any type.

Infrared pupillometry will be used to assess whether a painful stimulus results in pupillary reflex dilation (PRD). The extend of the PRD may be an indicator how painful a stimulus is. This may help to predict the amount of discomfort a patient will be experiencing after emergence from general anesthesia.

In addition to measuring the pupillary reflex dilation, we will also measure oscillations of pupil size before and after indiction of anesthesia, as well as during recovery. These spontaneously occuring oscillations in pupil size, also called hippus, appear to be sensitive to anesthetics and opioids. However, the effect of these drugs on hippus has not been systematically addressed.

The aim of the study is

1. to identify whether regional anesthesia techniques such as femoral and sciatic nerve blocks will block the PRD. This would allow assessment of block success in the anesthetized patient.
2. to correlate the extent of the pupillary reflex dilation and hippus in the anesthetized patient during and at the end of surgery with early postoperative pain scores and subsequent analgesia requirements. Such correlation would allow to predict the amount of postoperative pain before the patients emerge from general anesthesia.

DETAILED DESCRIPTION:
The planned study is a prospective cohort study.

Patients undergoing arthroscopic knee surgery of any type (debridements, repair of anterior (ACL) or posterior cruciform ligaments (PCL), meniscectomies, medial (MCL) or lateral collateral ligament (LCL) repair, as well as microfracture surgery will be enrolled.

During anesthesia, infrared pupillometry will be used to assess whether a painful stimulus results in pupillary reflex dilation (PRD). The extend of the PRD may be an indicator how painful a stimulus is. The PRD is measurable under general anesthesia in spite of the fact that the patient does not "feel" or experience the painful stimulus.

The aim of the study is

1. to identify whether regional anesthesia techniques such as femoral and sciatic nerve blocks (performed before the start of anesthesia) will block the PRD evoked by a painful stimulus such electrical stimulation before procedure start. This would allow assessment of block success in the anesthetized patient.
2. to correlate the extent of the pupillary reflex dilation and hippus in the anesthetized patient during and at the end of surgery with early postoperative pain scores and subsequent analgesia requirements. Such correlation would allow to predict the amount of postoperative pain before the patients emerge from general anesthesia.

Knee arthroscopies are routinely performed under general anesthesia with or without regional anesthesia, depending on the anticipated extent of surgery and the preferences of the anesthesiologist and surgeon. The assessment of the PRD and/or hipppus before emergence would identify those patients who would benefit from an additional nerve block before emergence to achieve better pain control immediately postoperatively and to reduce the demand for postoperative analgesics.

The planned investigation tries to achieve two novel findings. First, the measurement of the PRD at the start of surgery will demonstrate whether a nerve block successfully blocks the initial surgical stimulus. There is currently no method available that can assess block success in the anesthetized patient. Secondly, the measurement at the end of the surgery tries to predict the amount of pain following emergence from surgery. Pain may be experienced by patients without nerve blocks as well as with nerve blocks, as the latter may have failed or incomplete blocks, or may had a more extensive procedure that cannot be completely covered by the block administered preoperatively. Identifying these patients may allow treatment to minimize discomfort following emergence.

Pupillary reflex dilation describes the dilation of the pupil following a painful stimulus. The dilation last several seconds. Pupillometry using an infrared pupillometer allows the quantification of the reflex dilation. The PRD can be given a numerical value that reflects the extent of the dilation. A recently published study demonstrated the correlation of the extend of the PRD with pain scores and opioid requirements postoperatively. However, this study was done in awake patients following surgery. The aim of this study is to predict analgesia requirements in patients still under general anesthesia, before they experience postoperative pain. We expect that infrared pupillometry during general anesthesia can predict pain following surgery. Once this has been established, this knowledge and its application would allow the anesthesiologist to initiate pain-relieving interventions such as additional nerve blocks or administration of analgesics before emergence of the patients from general anesthesia.

In addition to measuring the pupillary reflex dilation, we will also measure oscillations of pupil size before and after induction of anesthesia, as well as during recovery. These spontaneously occurring oscillations in pupil size, also called hippus, appear to be sensitive to anesthetics and opioids. However, the effect of these drugs on hippus has not been systematically addressed.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years undergoing arthroscopic knee surgery of any type

Exclusion Criteria:

* Blindness
* Anisocoria
* History of opioid abuse
* Chronic pain patients
* Gastric Reflux Disease (due to the use of laryngeal masks in the study)
* Non english speaking patients
* Cognitive impairment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopedic Institute, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group: all enrolled patients undergo the same protocol/ treatment:
  Anesthesia Premedication, Induction and Maintenance Pupillometry after administration of anesthetic drugs
  Anesthesia Premedication, Induction and Maintenance: The enrolled patients receive standard of care general anesthesia for knee arthroscopy. No additional pharmacological interventions are performed in study participants.
  The administered drugs, as outlined in the arms section, are midazolam, fentanyl, propofol, and sevoflurane. Study patients receive analgesic drugs as needed in the recovery room if they experience pain.
  Pupillometry after administration of anesthetic drugs: All study patients receive the standard of anesthetic care. Every time a anesthetic drug has been administered, changes in pupillary oscillations will be recorded.
  Assessment of pupil size and movements by shining infrared light into the eye and measuring the reflection over a 20 s period
  The administered drugs are:
  Midazolam 1-2 mg
Period: Overall Study
Arm/Group | Intervention Group
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention Group
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Pain in Recovery Room
Description: Pain as assessed by visual analogue score at arrival of the patient in the recovery room Scale goes from 0-10, with 10 indicating the worst pain possible
Time Frame: at arrival in recovery room
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 24
score on a scale | 5 (2)

2. Secondary Outcome: Number of Patients we Were Able to Elicit a PLR Under Stable Experimental Conditions
Description: Pupillary Reflex Dilation is measured intraoperatively at incision and at the end of the case as a possible indicator of success of regional anesthesia.
  Measurement of this requires stable experimental conditions, most notably sufficient depth of anesthesia.
Time Frame: measurements were taken at two time points during surgery. Each measurement took 30 seconds
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 24
Participants | 0

3. Other Pre Specified Outcome: Hippus
Description: We assess the effects of various anesthetic drugs on pupillary unrest (hippus). More specifically, we record pupil diameters over 20 seconds and then perform a Fourier Analysis of the diameter changes. The endpoint variable is power of the oscillations over certain predefined frequency bins.
Time Frame: Before anesthesia start (baseline measurement) until discharge of the patient (on average 1-2 hours after arrival in the recovery room)
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Intervention Group
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

LIMITATIONS AND CAVEATS:
In patients under general anesthesia the PLR could not be seen with the stimulus chosen for the experiment. PLR recorded at the end of surgery were attributable to a lack of anesthesia. The trial was terminated after 24 subjects participated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No